CLINICAL TRIAL: NCT01721967
Title: Ranolazine for the Treatment of Angina in Hypertrophic Cardiomyopathy Investigation
Brief Title: Ranolazine for the Treatment of Chest Pain in HCM Patients
Acronym: RHYME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00039302; 3938381 (Other: Duke University)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: chest pain; dyspnea
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Chest Pain; Dyspnea | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranolazine (Experimental): Ranolazine, 500 mg for 60 days
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine
  Other Names: Ranexa

SUMMARY:
The purpose of RHYME is to evaluate the safety and efficacy of ranolazine in Hypertrophic Cardiomypathy patients with chest pain or dyspnea despite treatment with standard medical therapy. This is a small, pilot, open-label (non-randomized) study of an approved drug for the treatment of angina in a novel patient population (adult patient population with hypertrophic cardiomyopathy).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Left Ventricle wall thickness >/= 15mm in the absence of other condition causing hypertrophy
* Baseline Angina/Shortness of Breath Frequency of > 2 episodes per week
* Willing to provide informed consent

Exclusion Criteria:

* Severe stenotic valvular disease
* Severe valvular regurgitation except mitral regurgitation due to systolic anterior motion
* Significant (>60% stenosis) coronary artery disease
* Acute coronary syndrome within 30 days
* Severe heart failure defined as LV systolic dysfunction with Ejection Fraction <40% or NYHA class 4 symptoms
* Severe renal impairment (glomerular filtration rate, <30 mL/min/1.73 m2)
* Moderate-severe hepatic impairment (Child-Pugh classes B and C)
* Hospitalization for cardiac reason within 3 months of enrollment
* Anticipated changes to treatment of HCM within study period, including medications, device implantation, or septal reduction therapies
* Concomitant use of ketoconazole, macrolide antibiotics, and HIV protease inhibitors
* Active myocarditis, pericarditis, or restrictive cardiomyopathy
* Non-cardiac terminal illness with expected survival less than 6 months
* Women who are of childbearing potential
* Inability to perform or adhere to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ranolazine
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Seattle Angina Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The SAQ is a self-report instrument with 19 items that yields five subscale scores: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life.
  units on a scale
    Physical limitation | 49.6 (18.7)
    Anginal stability | 45.5 (27.0)
    Anginal frequency | 65.5 (13.4)
    Treatment satisfaction | 85.2 (12.6)
    Quality of life | 40.9 (24.6)
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: units on a scale] — Similarly, the Kansas City Cardiomyopathy Questionnaire (KCCQ) is a new, self-administered, 23-item questionnaire developed to provide a better description of health-related quality of life in patients with heart failure. It quantifies, in a disease-specific fashion, physical limitation, symptoms (frequency, severity and recent change over time), quality of life, social interference and self-efficacy. All categories of questions are scored from 0-100, with higher number indicating better health.
  units on a scale
    Physical limitation | 61.7 (20.6)
    Symptom stability | 43.2 (16.2)
    Symptom frequency | 56.4 (20.6)
    Symptom burden | 55.3 (29.4)
    Total symptom score | 55.9 (24.2)
    Self-efficacy | 78.4 (21.7)
    Quality of life | 39.4 (26.6)
    Social limitation | 46.0 (31.5)
    Overall summary | 51.2 (22.3)
    Clinical summary | 58.8 (20.9)

OUTCOME MEASURES:

1. Primary Outcome: QT Interval
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Ranolazine
Number analyzed (Participants) | 11
msec | 462.8 (27.4)

2. Primary Outcome: Number of Adverse Events Considered Probably or Possibly Related to Study Drug
Description: Number of events that are considered probably or possibly related to study drug.
Time Frame: 60 Days
Measure: Number; unit: adverse event
Arm/Group | Ranolazine
Number analyzed (Participants) | 14
adverse event | 10

3. Primary Outcome: Drug Tolerability
Description: Total number of patients that tolerated 1,000mg BID dose and 500 mg BID dose
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Ranolazine
Number analyzed (Participants) | 14
participants
  1000 mg BID | 9
  500 mg BID | 4

4. Secondary Outcome: Improvement in Number of Episodes of Angina Per Week
Description: Efficacy of ranolazine in HCM patients with respect to improvements in angina frequency (number of episodes of angina per week).
Time Frame: Baseline and 60 Days post treatment
Population: episodes of angina per week was not collected
Arm/Group | Ranolazine
Number analyzed (Participants) | 0

5. Secondary Outcome: Seattle Angina Questionnaire (SAQ)
Description: The Seattle Angina Questionnaire (SAQ) is a self-administered, 19-item questionnaire, a cardiac disease-related quality-of-life measure. The SAQ is well validated and sensitive to clinical changes. It has five subscales: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life.
Time Frame: 60 Days post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranolazine
Number analyzed (Participants) | 11
units on a scale
  Physical limitation | 61.4 (18)
  Anginal stability | 90.0 (21.1)
  Anginal frequency | 86.0 (12.7)
  Treatment satisfaction | 90.6 (11.5)
  Quality of life | 70.8 (11.3)

6. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ) (scores range from 0 to 100 with higher scores representative of a higher quality of life; clinically important changes are considered > 10 points and >5 points, respectively, as previously established
Time Frame: 60 days post treatement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranolazine
Number analyzed (Participants) | 11
units on a scale
  Physical limitation | 72 (20.6)
  Symptom stability | 72.7 (26.1)
  Symptom frequency | 72.2 (20)
  Symptom burden | 75 (24.2)
  Total symptom score | 73.6 (21.3)
  Self-efficacy | 85.2 (14.6)
  Quality of life | 65.2 (25.8)
  Social limitation | 66.1 (31.2)
  Overall summary | 69.8 (23.5)
  Clinical summary | 74 (20.5)

ADVERSE EVENTS:
Arm/Group | Ranolazine
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=14)
Leg Weakness (Musculoskeletal and connective tissue disorders) | 1
dizziness (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes